CLINICAL TRIAL: NCT04199013
Title: Comparison of Ropivacaine With or Without Fentanyl in Spinal Anaesthesia for Lower Limb Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, ABINASH DHOJ JOSHI, RESIDENT DOCTOR, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 125/(6-11)E2/076/077
Record Dates: First submitted 2019-12-06; First posted 2019-12-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Leg Injury; Arthroplasty, Replacement, Knee
Keywords: 0.75% ROPIVACAINE; FENTANYL; SPINAL ANAESTHESIA
MeSH Terms: conditions — Leg Injuries | interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine With Fentanyl (Active Comparator): 2.5ml of 0.75% Isobaric ropivacaine with 0.5ml (25mcg) Fentanyl
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution; Drug: Fentanyl Citrate
- Ropivacaine Without Fentanyl (Active Comparator): 2.5ml of 0.75% Isobaric Ropivacaine with 0.5ml of Normal Saline
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.75% Injectable Solution — Patients in Group R will receive subarachnoid injection of 2.5 ml of 0.75% isobaric ropivacaine (18.75 mg) and 0.5 ml normal saline while patients in Group RF will receive subarachnoid injection of 2.5 ml 0.75% of isobaric ropivacaine (18.75 mg) and 0.5 ml fentanyl (25 μg).
  Other Names: ROPIN 0.75%
Drug: Fentanyl Citrate — Patients in Group R will receive subarachnoid injection of 2.5 ml of 0.75% isobaric ropivacaine (18.75 mg) and 0.5 ml normal saline while patients in Group RF will receive subarachnoid injection of 2.5 ml 0.75% of isobaric ropivacaine (18.75 mg) and 0.5 ml fentanyl (25 μg).
  Other Names: FENTYL
  Arms: Ropivacaine With Fentanyl

SUMMARY:
There has been a wide variety of use of anaesthetic agents along with adjuncts during subarachnoid block. The quest for attaining adequate analgesia and anaesthesia has always been shadowed by the concurrent deleterious effect of the anaesthetic agent. Ropivacaine as an anesthetic agent has proven to meet the desired goals of anaesthesia while minimizing the potential side effects. The addition of different adjuncts has shown to enhance the analgesic property, prolong the duration of sensory blockade and decrease the dose related adverse effects of the local anaesthetics. Fentanyl in this regards has also shown some promising effects. Thus we compare the use of ropivcaine as a single agent versus ropivacaine along with an adjunct (Fentanyl) to attain the desired anesthetic effect while minimizing the associated side effects.

DETAILED DESCRIPTION:
Spinal anaesthesia has been a widely used mode of anaesthesia for lower abdominal and extremity surgeries. It blunts the "stress response" to surgery, decreases intraoperative blood loss, lowers the incidence of postoperative thromboembolic events, and decreases the morbidity in high-risk surgical patients. It serves as a useful method to extend analgesia into the postoperative period, where its use has been shown to provide better analgesia than parenteral opioids. In order to improve further and understand safety issues as well as the clinical use of spinal anesthesia, new local anesthetics and analgesic additives are being investigated for different application. With patient safety and comfort being the ultimate goal of any health practice, one must keep in mind about the side effects and related concerns of spinal anesthesia while achieving the desired level of anaesthesia and analgesia. Adequate anesthesia and analgesia during and post-surgery along with early ambulation and discharge seems to be the perfect recipe for the conduction of spinal anaesthesia in the current practice. Ropivacaine is one local anesthetic that could have the potential in this area. Ropivacaine is an amide local anesthetic with properties similar to bupivacaine producing similar sensory block at equipotent doses, but with a shorter duration of motor block. Thus, ropivacaine has a greater degree of motor sensory differentiation, which could be useful when motor blockade is undesirable. Ropivacaine blocks nerve fibers involved in pain transmission (A∂and C fibers) to a greater degree than those controlling motor function (Aβ fibers).Blockade of Aα and Aβ is slow and hence produces lesser motor blockade than bupivacaine. Though 40-50% less potent than bupivacaine, ropivacaine in an equipotent ratio of 1.5:1 produces results in a similar clinical profile with good preservation of motor function. Hence, its shorter duration, faster recovery of motor function, lower toxicity profile, and minimal hemodynamic alterations have been identified as a potential benefit for surgery of intermediate duration as well as for ambulatory surgery.

Though the use of bupivacaine is widespread, ropivacaine in the recent times has been used as a spinal anaesthetic agent and evaluated in many procedures because of its equivalent spinal anaesthetic effect and its lower risk of neurotoxicity and cardiotoxicity, compared with bupivacaine. In addition, there have been reports of fatal cardiovascular toxicity following use of bupivacaine in regional anesthesia.

Subarachnoid opioids with local anesthetics have become a well-accepted practice in spinal anesthesia for surgical procedures. Several combinations of local anesthetics such as lidocaine, bupivacaine, or ropivacaine, and opioids such as fentanyl have been reported for a variety of surgical procedures. The addition of small-dose fentanyl (10-25 μg) intrathecally to local anesthetics during spinal anesthesia has been shown to enhance duration of sensory analgesia.The addition of adjuvants to ropivacaine has shown to improve the quality of intra-operative and postoperative analgesia without compromising its benefits such as early mobilization and early voiding. Parlow et al. established the fact that hypobaricity influenced the extent of subarachnoid block and explained high cephalic levels of sensory block when fentanyl was added to isobaric local anesthetic solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for lower limb surgeries under spinal anaesthesia.

Exclusion Criteria:

* Patient refusal. Patient height less than 150 cm. History of hypersensitivity to study drugs. Pregnancy. Patient unable to communicate verbally.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time for block regression to S2 segment | Up till 5 hours from spinal block
  The total duration of sensory blockade will be defined as the time interval between spinal anesthesia till block regression to S2 segment. Time for block regression to S2 segment will be noted every 30 mins after end of surgery.

SECONDARY OUTCOMES:
Total duration of analgesia | Uptill 12 hour post surgery
  Duration of analgesia will be defined as time interval from subarachnoid injection to the point where patients demanded rescue analgesics for pain relief. Analgesia for pain management will be given as per the hospital protocol.

CONTACTS AND LOCATIONS:
Overall Officials: ANIL SHRESTHA, MD, Study Chair — TRIBHUVAN UNIVERSITY TEACHING HOSPITAL
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No